CLINICAL TRIAL: NCT00822614
Title: The Safety of Fentanyl TAIFUN Treatment After Titrated Dose Administration and the Current Breakthrough Pain Treatment for Breakthrough Pain in Cancer Patients
Brief Title: Safety of Fentanyl TAIFUN Treatment
Acronym: FINDS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akela Pharma, Inc. (Industry)
Responsible Party: Elvi Metsaranta, Akela Pharma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL_700_014
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Breakthrough Cancer Pain
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — Analgesics, Opioid; Morphine; Hydromorphone; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator (Active Comparator): Current BTP Medication
  Interventions: Drug: Opioid
- Fentanyl TAIFUN (Experimental): Titration for dose confirmation followed by observation period
  Interventions: Drug: Fentanyl TAIFUN

INTERVENTIONS:
Drug: Fentanyl TAIFUN — Inhalation of Fentanyl via TAIFUN inhaler
  Arms: Fentanyl TAIFUN
Drug: Opioid — Current optimized BTP treatment
  Other Names: Fentanyl transdermal; Morphine Sulfate; Hydromorphone; Oxycodone
  Arms: Active Comparator

SUMMARY:
A Multicenter, Multinational, Randomized, Open-Label, Parallel-Group Trial to Evaluate hte Safety of Fentanyl TAIFUN Treatment after titrated Dose Administration and the Current Breakthrough Pain Treatment for Breakthrough Pain in Cancer Patients on Maintenance Opioid Therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 18 Years or older
* A medically documented diagnosis of cancer
* Use of a fixed round the clock dose of opioid as maintenance therapy with a dose equivalence of at least 60mg of oral morphine/ day, or at least 25 mcg of transdermal fentanyl/ hour, or at least 30 mg of oral oxycodone daily, or at least 8 mg of oral hydromorphone daily. Current opioid treatment for at least 7 days prior to randomization
* Current use of opioid medication for BTP
* At least 4 episodes of BTP per week, with peak intensity of at least 4 on the NPS at pain onset. No more than 4 BTP episodes per day.
* PIFR of at least 20L/min
* Karofsky Performance Status of 40 or better
* Life expectancy of at least 12 weeks
* Written Informed Consent

Exclusion Criteria:

* Uncontrolled or rapidly increasing BTP
* Symptomatic intracranial tumors or cerebral metastases
* Persistent symptomatic asthma
* Patients unable to use the inhaler
* Inadequate lung function, as defined by PEFR <60%
* Hypersensitivities, allergies or contraindications to fentanyl or the study medication components
* A recent history of alcohol or substance abuse (in the past 1 year)
* Radiotherapy to the thorax within 30 days of the beginning of the titration phase
* Cognitive impairment or any neurological of psychiatric disease which could compromise the ability of the patient to complete the assessments
* Participation in any clinical study with an experimental drug within 30 days of randomization
* Any clinical condition or medical history which, in the opinion of the investigator would not allow for the safe completion of the study or the safe administration of the study drug
* Pre-menopausal women who are not surgically sterile and/or have a positive pregnancy test at baseline visit and/ or are of child bearing potential and are not using a reliable method of birth control or do not plan to continue using this method throughout the study and/or who are nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
AE Profile | 28 Days
To characterize the safety of Fentanyl TAIFUN treatment vs. the current BTP treatment based on the AE profile | 28 days

SECONDARY OUTCOMES:
To estimate the proportion of patients taht can be titrated to an effective dose of Fentanyl TAIFUN | 28 Days
To evaluate the efficacy of Fentanyl TAIFUN with the titrated dose and the current BTP treatment with the confirmed dose | 28 Days
To evaluate patients's preference between Fentanyl TAIFUN and the baseline BTP medication | 28 Days
To evaluate the sustained analgesic effect of Fentanyl TAIFUN and the current BTP treatment | 28 Days

CONTACTS AND LOCATIONS:
Locations (1):
- NZOZ, Włocławek, Wolnosc, Poland